CLINICAL TRIAL: NCT06896864
Title: Cochlear Implantation in Assiut University Hospital Experience
Brief Title: Cochlear Implantation Experience
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Sayed Hussein, cochlear implantation in Assiut university hospital experience, Assiut University
Other Study IDs: CI experience
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cochlear Function Disorder
MeSH Terms: interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: cochlear implantation — After the surgery, patients typically undergo a period of recovery and healing. several factors including age at implantation, pre- and post-operative therapy, and parental involvement

SUMMARY:
Evaluating the effectiveness and outcomes of cochlear implants in individuals with hearing loss,identifying common complications or risks associated with cochlear implantation, including device failure, surgical complications, or issues related to the patient's anatomy

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe to profound bilateral sensorineural hearing loss who were candidates for CI.

Patients who regularly use their cochlear implant device as recommended.

Exclusion Criteria:

* Non-Sensorineural Hearing Loss - Non-Functional Auditory Nerve - . Severe Mental or Cognitive Impairments

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All cases implanted between 2014-2024 Patients who regularly use their cochlear implant device as recommended.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-04-08 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Post-Surgical Complication Rate: Infection, device failure,Measures auditory progression | Baseline